CLINICAL TRIAL: NCT04282343
Title: A Phase 2 Trial of the Discussion of Cost (DISCO) App as an Intervention to Improve Financial Outcomes in Hematologic Cancer Patients
Brief Title: DISCO Application for the Improvement of Financial Outcomes in Patients With Hematologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Lauren Hamel, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2019-131
Record Dates: First submitted 2020-02-09; First posted 2020-02-24 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Plasma Cell Myeloma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Patients are randomized to 1 of 2 arms: ARM I: Patients receive usual care consisting of general cancer treatment information on a sheet of paper before attending video-recorded meetings with their oncologist to discuss treatment plan; or ARM II: Patients use the DISCO education and communication app before attending video-recorded meetings with their oncologist to discuss treatment plans. After completion of study, patients are followed up at 3 months.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Trained research assistants and oncologists
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I- Usual care (Other): Patients receive usual care consisting of general cancer treatment information on a sheet of paper before attending video-recorded meetings with their oncologist to discuss treatment plans.
  Interventions: Behavioral: Usual Care
- Arm II - DISCO app (Other): Patients use the DISCO education and communication app before attending video-recorded meetings with their oncologist to discuss treatment plans.
  Interventions: Behavioral: The DISCO App

INTERVENTIONS:
Behavioral: The DISCO App — Patients will receive an individually-tailorable cancer treatment cost education and communication intervention delivered on an iPad just prior to meeting with their oncologist.
  Arms: Arm II - DISCO app
Behavioral: Usual Care — Patients randomized to this arm will receive usual care.
  Arms: Arm I- Usual care

SUMMARY:
This phase II trial studies how well the DIScussion of COst (DISCO) application (app) works in improving financial outcomes in patients with hematologic cancer. The DISCO app is an electronic, highly scalable and tailorable education and communication intervention that may help researchers learn more about improving how patients and oncologists discuss cancer treatment costs

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the effectiveness of the DISCO app on prompting patient-oncologist treatment cost discussions during patient-physician interactions (as observed in video recordings), patient outcomes related to financial toxicity immediately after the patient-oncologist interaction, and at a 3-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* ONCOLOGISTS: Eligible if they treat patients with chronic lymphocytic leukemia (CLL), chronic myelogenous leukemia (CML), or multiple myeloma (MM) cancers
* PATIENTS: Able to read and write in English
* PATIENTS: Have a confirmed diagnosis of CLL, CML, or MM cancers
* PATIENTS: Are scheduled to see an oncologist at Karmanos Cancer Institute (KCI) Detroit or KCI Farmington Hills/Weisberg for an initial or change in treatment discussion

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Presence of cost discussion observed via video recordings of patient-physician treatment discussions. | Observed during the video-recorded patient-physician interaction.
  Number of participates who have a treatment cost discussion will be evaluated with a validated observational scale. This is an investigator-developed scale and its called the Discussion of Cost (DISCO) scale. A higher score means a better outcome.

SECONDARY OUTCOMES:
Referrals for financial or psychological support | Immediately after the patient-physician interaction
  Number of participants who receive a referral for financial or psychological support will be evaluated with a self-report item. This an investigator-developed yes/no one-item response. A "yes" response is a better outcome than a "no" response.
Self-efficacy in managing treatment cost | Immediately after the patient-physician interaction
  How efficacious each participant feels about managing treatment costs will be evaluated with an adapted validated self-report scale and its title is: Managing Treatment Cost Self-Efficacy scale. This an investigator-adapted scale, and a higher score means a better outcome (max =7; min = 1).
Self-efficacy in patient-physician interactions | Immediately after the patient-physician interaction
  How efficacious each participant feels about interacting with physicians will be evaluated with a validated self-report scale, and its title is: Perceived efficacy in patient-physician interactions (PEPPI). A higher score means a better outcome.(max =50; min = 10)
Treatment cost distress | Immediately after the patient-physician interaction
  How distress each participant feels about how much their treatment will cost them will be evaluated with an investigator-developed validated self-report scale, and its title is: Treatment Cost Distress Scale. A higher score means a worse outcome. (max =7; min = 1)
Anticipated material hardship | Immediately after the patient-physician interaction
  How much anticipated material hardship each participant feels they may experienced due to treatment costs will be evaluated with a validated self-report scale, and its title is: Economic Hardship Scale. A higher score means a worse outcome. (max =7; min = 1)
Financial toxicity | 3 months after the patient-physician interaction
  How much material and psychological hardship the patients experiences due to treatment cost will be evaluated with a validated self-report scale, and its title is: Comprehensive Score for Financial Toxicity (COST). A higher score means a worse outcomes. (max=7; min=1)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Hamel, PhD, Principal Investigator — Barbara Ann Karmanos Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No